CLINICAL TRIAL: NCT06174740
Title: Neural Correlates of Multisensory Stimulation in Healthy Older Adults
Brief Title: Brain Imaging and Behavioural Changes Following Cued-movement Training of Finger Sequences in Healthy Older Adults
Acronym: NMSOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, Rebecca Schaefer, Associate Professor, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-08-23-RS Schaefer-V2-4097
Record Dates: First submitted 2023-06-21; First posted 2023-12-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Aging; Music; Motor Activity; Magnetic Resonance Imaging; Neuronal Plasticity
Keywords: auditory; multisensory; stimulation; auditory cued; music based; music therapy training; rhythmic auditory stimulation; Diffusion Magnetic Resonance Imaging; Diffusion Tensor Imaging; motor learning; movement training
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either the audiovisual condition (Experimental Group) or visual cues only condition (Control Group). A randomization list stratified by gender will be generated before commencing data collection.
Who Masked: Outcomes Assessor
Masking Description: The order of the allocation for new inclusions will be concealed from the assessors. Researchers administering assessments at the two time points will be masked and concealed from the randomization and participant allocation. Researchers involved in the MRI acquisition and analysis will collect the data under a different participant identifier (ID) than the ID used to conduct MRI analysis, and will follow an analysis script designed before data collection is completed, where applicable. Participants, and researchers may not be masked from the conditions due to practical reasons relating to the presence of auditory stimuli in the same or nearby vicinity, or interacting with the participants regarding the presence of auditory stimuli, which is the main intervention being investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music-Cued Audiovisual Motor Training (Experimental): Participants will be instructed on the task which they will perform at home online using a keyboard. The training involved auditory-cued audiovisual finger movement sequence learning task. Participants will complete an online computer-based training of 20 minutes at home 3 times per week for the duration of 8 weeks, and a total of 24 sessions, the duration and number of sessions.
  Interventions: Behavioral: Music-cued audiovisual motor training
- Visually-Cued Motor Training (Active Comparator): Participants will be instructed on the task which they will perform at home online using a keyboard. The training involved visual cues for finger-movement sequence learning task. Participants will complete an online computer-based training of 20 minutes at home 3 times per week for the duration of 8 weeks, and a total of 24 sessions, the duration and number of sessions
  Interventions: Behavioral: Visually-cued motor training

INTERVENTIONS:
Behavioral: Music-cued audiovisual motor training — In addition to visual cues, music stimuli guide finger sequence movement both rhythmically (temporal component) and sonically (pitch-finger alignment).
  Other Names: music-based training; music-cued training; music-based motor learning; multisensory stimulation; rhythmic auditory stimulation
  Arms: Music-Cued Audiovisual Motor Training
Behavioral: Visually-cued motor training — Visual cues guide finger sequence movement by indicating which finger to move in alignment with the position and of the visual cue.
  Other Names: Control Group
  Arms: Visually-Cued Motor Training

SUMMARY:
The goal of this study is to examine changes in the brain, behavior, and personal experience when music is used to guide learning of finger movement sequences (compared to visual stimuli alone) in healthy older adults. The main research questions this study aims to answer are:

1. Is auditory-based motor training associated with increased structural integrity of brain white matter tracts (connecting auditory-motor regions) compared to motor training with visual cues only?
2. Is auditory-based motor training (as compared to visual clues only) associated with increased brain cortical thickness, and changes in brain activation while performing a task in the MRI and while at rest, in auditory and sensorimotor regions?
3. Does auditory-based motor training lead to greater motor improvement on the trained task compared to a visually cued motor training?
4. Does auditory-based motor training lead to greater improvement on thinking, movement, and self-reported wellbeing measures, compared to visual cues alone?

In an 8-week home training, participants will be randomized into either the music-cued motor learning (Experimental Group) or visually cued only condition (Control Group), participants will complete the following measures before-and-after the training is administered at week 1 and in the end of the 8-week trial:

* MRI scans (structural and functional)
* Behavioral measures (motor, cognition)
* Questionnaires administered pre-and-post training (psychosocial functioning).
* Questionnaires administered once only (personality traits, musical background)
* In between measures, participants will follow an online computer-based training at home of 20 minutes per session, 3 times per week for 8 weeks, for a total of 24 sessions constituting 8 hours of training.

DETAILED DESCRIPTION:
Rationale: Music interventions targeting motor recovery are increasingly used in clinical settings with motorically impaired patients. In recent years, research started to demonstrate the mechanism underlying motor recovery by moving to music. While neuroimaging studies began to elucidate the neural correlates of music-based movement, most of these studies have been conducted on young adults, whereas the average age at onset of movement disorders which are the target of music therapy is in the 6th decade of life. Therefore, in this study the investigators aim to elucidate the underlying mechanisms of music-based movement in healthy older adults using a motor learning, finger sequence task to a musical rhythm. The results of the study have implications for motor learning with music in the aging person and neural plasticity in old age, and may reveal the benefit of adding music-cues to motor activities for motor, cognitive, and motivational outcomes in older adults.

Objective: The goal of the current study is to examine structural and functional neural correlates, as well as changes in behavioral and self-report measures of audiovisual music-based motor training compared to an identical motor training using visual cues only. The study focuses on white matter changes as the primary objective as the researchers are interested in connections between auditory and motor brain regions implicated in music-cued motor training. The research will examine brain activation, and changes in grey matter volume as secondary neuroimaging outcomes. Moreover, the study will also examine improvement on the trained task (outside of the MRI scanner), and changes on standardized measures of motor and cognitive function, as well as self-report measures of psychological wellbeing.

The main hypothesis is that the music-based motor training group will show greater white matter integrity of the arcuate fasciculus and greater density of cortical thickness in motor areas in the right brain hemisphere opposite to the trained left hand, as well as greater changes in brain activation while performing the task and at rest. The music group is expected to show greater improvement on the trained task, and measures of motor and cognitive function, as well as self-report measures of wellbeing (motivational, mood, and experience). As an exploratory measure, the study will assess changes in dual-task interference before and after the training as a far-transfer measure of the training, both in motor function and the underlying brain function.

Study design: In an 8-week longitudinal between-group design, participants will be randomized into two groups and will participate in pre-and-post MRI scans and behavioral measures, administered at baseline (week 1) and end of trial (week 8). The learning of an audio-visual finger movement sequence task will be compared to training on the same motor sequence with visual cues only. Participants will be assessed before and after the 8-week training on MRI and behavioral measures.

Study population: A total of 50 healthy older adults (60 years and older) will be recruited for this study and randomized into two groups of 25 participants each. Inclusion criteria are being right-handed (assessed by the Edinburgh Handedness Inventory), neurologically and physically healthy adult aged 60 or older (a previous diagnosis of a neurological/psychiatric illness that is symptom-free and for which no treatment was necessary for at least 5 years may be included), other physical health conditions that are stable (no change in diagnosis or treatment in the past 2 years may be included), having age-normal cognitive function (as assessed by a score of ≥24 on the MMSE), age appropriate normal or corrected vision and hearing ability, speaking fluent Dutch, and not currently receiving musical training. Participants should have access to a computer to complete the training at home. Participants will be recruited through various channels in the Netherlands including ageing organizations, (social) media, and study recruitment websites.

Sample Size: In a previous study with a longitudinal design using the same learning task in healthy young adults, the researchers found a medium size effect for changes in white matter tracts connecting auditory and motor regions (i.e., arcuate fasciculus) in the brain hemisphere opposite the trained hand. Therefore, it is estimated that the sample size needed to show a similar medium sized effect would be 22 per group, however, this number is increased to 25 healthy older participants per group to account for additional drop out at the analysis stage.

Intervention: Two groups will receive a similar intervention of finger sequence movement learning following visual cues with (or without) rhythmic auditory stimulation. Participants will be trained on the task at the laboratory before baseline measures. Participants will continue training at home online on a computer and keyboard for 20 minutes per session 3 times per week for 8 weeks for a total of 24 sessions. The Music group will train the finger sequence with the aid of visual cues in synchrony with a musical rhythm, while the Control group will receive the same visual stimulation with no auditory component.

Main study parameters/endpoints: The main parameter is change in white matter tracts underlying auditory-motor regions (arcuate fasciculus) in the brain hemisphere opposite the trained hand, contrasting before and after training, and between hemispheres. Secondary MRI parameters focus on cortical thickness changes in primary, premotor, and supplementary motor areas, task-related brain activation in the premotor cortex, and resting-state functional connectivity of auditory-motor regions. Motor performance on the cued motor sequence task will be assessed by measuring the accuracy of the key presses and the timing stability in synchrony with the onset of the cue. Changes in the scores of standardized motor and cognitive measures, and self-reported questionnaires on motivational and mood indices will be compared between groups and timepoints. As an exploratory outcome, the study will also assess changes in dual-task interference before and after the training both behaviorally and in terms of associated brain activity while performing the task.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (assessed by the Edinburgh Handedness Inventory),
* Neurologically and physically healthy adults (a previous diagnosis of a neurological/psychiatric illness that is symptom-free and for which no treatment was necessary for at least 5 years may be included), other physical health conditions that are stable (no change in diagnosis or medication in the past 2 years may be included)
* aged 60 or older,
* Age-normal cognitive function (as assessed by a score of ≥24 on the MMSE),
* Age appropriate normal or corrected vision and hearing ability,
* Speaking fluent Dutch,
* Not currently receiving musical training.
* Participants should have access to a computer and internet to complete the training at home.

Exclusion Criteria:

* MRI contraindications (e.g., having ferromagnetic metals, such as implants, or claustrophobia)
* Starting or currently engaged in hand training, including musical training, and for example knitting, type-writing, or other hobbies (musical activities such as dancing or singing that do not involve the hand).
* Changes in medications that may affect fMRI measures.
* Not being able to follow the training at the laboratory or at home, or not completing the practice at home despite alerts and reminders.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in white matter diffusivity of the arcuate fasciculus | Baseline and week 8
  Change to white matter diffusivity (baseline to post training; within and between hemispheres contralateral to the trained vs. untrained hand) will be assessed by comparing fractional anisotropy (FA) radial diffusivity (RD), and mean diffusivity (MD) of the left and right arcuate fasciculus between groups across the two timepoints, pre-and post-training in the hemisphere contralateral to the trained hand, and between the hemispheres.

SECONDARY OUTCOMES:
Change in cortical thickness in motor areas from baseline at week 8 | Baseline and week 8
  Change from baseline in cortical thickness of the primary, premotor, and supplementary motor areas contralateral to the trained hand before and after training will be compared between the musical group and the control group focusing on regions of interest in sensorimotor areas. Cortical thickness is measured using an initial surface generated for each hemisphere by tiling the outside of the white matter mass for that hemisphere. This initial surface is then refined to follow the intensity gradients between the white and gray matter (this is referred to as the white surface). The white surface is then nudged to follow the intensity gradients between the gray matter and cerebrospinal fluid (this is the pial surface). The white and pial surfaces are overlaid on the original T1-weighed image, and the distance between the white and the pial surfaces is measured to determine the thickness at each location of cortex.
Change form baseline in task-based functional magnetic resonance imaging (fMRI) activation in the premotor cortex at week 8 | Baseline and week 8
  Change from baseline in task-based functional MRI activation (Blood Oxygen Level Dependent; BOLD) in the premotor cortex, examining the contrast (Cued Tapping vs Rest) at week 8.
Change from baseline in resting state fMRI connectivity in the auditory and sensorimotor networks at week 8 | Baseline and week 8
  Change from baseline in resting state connectivity will focus on nodes of auditory network and sensorimotor network strength in functional MRI activation at week 8
Motor performance on the cued motor sequence task across three time points (pre-post measurement visits, and mid-trial online) based on accuracy of the key presses | Baseline, week 4, and week 8
  Motor performance on the cued motor sequence task across three time points (pre-post measurement visits of the 8-week training, and mid-trial at week 4 online) based on accuracy of the key presses. The number of correctly performed motor sequences and movement will be averaged for trained and untrained sequences.
Motor performance on the cued motor sequence task across three time points (pre-post measurement visits, and mid-trial online) based on the timing stability and synchrony with the onset of the cue. | Baseline, week 4, and week 8
  Motor performance on the cued motor sequence task across three time points (pre-post measurement visits of the 8 week training, and mid-trial at week 4 online) based on the timing stability in synchrony with the onset of the cue. The number of correctly performed motor sequences and movement will be averaged.
Change from baseline in the scores of Grooved Pegboard Task at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Grooved Pegboard Task (measured in time in seconds) for both the dominant and non-dominant hand. A total of 240 seconds is the maximum allowed (minimum of 0), where a higher score indicates worse outcome.
Change from baseline in the scores of Box and Blocks Test at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Box and Block test (measured in number of blocks transferred in one minute, rule breaks are deducted) for both the dominant and non-dominant hand. A score of 150 is the maximum (minimum of 0), where a higher score indicates a better outcome.
Change from baseline in the scores of Digit Span Forward at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Digit Span task (number of correctly recalled digits in a sequence is recorded), a maximum score of 2-9, with a higher score meaning a better outcome.
Change from baseline in the scores of Digit Span Backwards at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Digit Span task (number of correctly recalled digits in a sequence is recorded) with a score ranging from 2-8 and a higher score indicating better outcome.
Change from baseline in the scores of Trail Making Test at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Trail Making Test (measured in time over 5 trials). The final score is trial 4 (letter-switching) (score range: 0-240) minus the average of trials 1,2, 3, and 5 (Visual scanning, number sequencing, letter sequencing, and motor speed, respectively). The minimum possible score is 0 and the maximum is 240, where a higher score indicates a worse outcome.
Change from baseline in the scores of Stroop Color Word Interference Test at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Stroop Color Word Interference Test (the combined time during the two congruent trials is subtracted from the time during the non-congruent trial), the lowest possible score is 0 and the maximum is 180, where a higher score indicates a worse outcome.
Change from baseline in the scores of Verbal Fluency Test at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Verbal Fluency Test (total number of correct responses across trials excluding repeats, and deducting errors for phonemic and categorical subtests are recorded), where a higher score indicates better performance, a minimum of 0 and a maximum of 480.
Change from baseline in the scores of Rey Auditory Verbal-Learning Test at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Rey Auditory Verbal-Learning Test, the number of correct responses is recorded for both immediate, interference and delayed recall trials, the final score is the highest achieved number on the learning trails (0 - 15) minus the delayed recall score (0 - 15), where a higher score indicates a worse outcome. The maximum score is 15 and the lowest is -15.
Change from baseline in scores of Quality of Life measure at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the EuroQol- 5 (Dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression) range from 1-5 where a higher number is a worse outcome, and a visual analogue scale from 0-100 where a higher number is a better outcome.
Change from baseline in scores of mood measure at week 8 | Baseline and week 8
  Change from baseline to week 8 in scores of the Depression Anxiety Stress Scale, where Depression symptoms related items: 3, 5, 10, 13, 16, 17, 21 (range from 0-21) Anxiety disorder-related items: 2, 4, 7, 9, 15, 19, 20 (range from 0-21) Stress-related items: 1, 6, 8, 11, 12, 14, 18 (range from 0-21), where a higher score indicates a worse outcome for all domains.

OTHER OUTCOMES:
Change from baseline in brain activation during a dual cognitive-motor interference task at week 8 | Baseline and week 8
  Change from baseline to week 8 in brain activation during a dual cognitive-motor interference task at week 8. Participants are asked to conduct a finger tapping task, and a letter counting task separately (Single Task condition), and a third trial in which participants are asked to perform both tasks simultaneously (Dual Task condition), fMRI cortical activation will be compared at baseline and at week 8 by canceling the role of the single tasks from the dual task, and comparing the two groups.
Change from baseline in performance of dual cognitive-motor interference task at week 8 | Baseline and week 8
  Change from baseline to week 8 in performance of the dual cognitive-motor interference task at week 8. Participants are asked to conduct a finger tapping task, and a letter counting task separately (Single Task condition), and a third trial in which participants are asked to perform both tasks simultaneously (Dual Task condition). Scores on the task will be compared at baseline and at week 8 by contrasting the role of the single tasks from the dual task and quantifying any decreases/interference related to the dual task, and comparing the two groups.
Changes from baseline in white matter diffusivity of the corticospinal tract at week 8 | Baseline and week 8
  Changes (baseline to post training; within and between hemispheres contralateral to the trained vs. untrained hand) comparing fractional anisotropy, radial diffusivity, and mean diffusivity of the corticospinal tract between groups across the two timepoints, pre-and post-training in the hemisphere contralateral to the trained hand, and between the hemispheres.
Change from baseline in associations between cognitive and white matter diffusivity measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test), and self-report measures and trained tasks) and MRI changes in white matter diffusivity (as measured by fractional anisotropy of the left arcuate fasciculus measures) at baseline and at week 8.
Change from baseline in associations between motor measures and white matter diffusivity measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test) and MRI changes in white matter diffusivity (as measured by fractional anisotropy of the left arcuate fasciculus measures) at baseline and at week 8.
Change from baseline in associations between self-report measures and white matter diffusivity measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number)) and MRI changes in white matter diffusivity (as measured by fractional anisotropy of the left arcuate fasciculus measures) at baseline and at week 8.
Change from baseline in associations between motor training performance and white matter diffusivity measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue) and MRI changes in white matter diffusivity (as measured by fractional anisotropy of the left arcuate fasciculus measures) at baseline and at week 8.
Change from baseline in associations between cognitive measures and cortical thickness measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test), and self-report measures and trained tasks) and MRI changes in cortical thickness (measured as the distance between the white and the pial surfaces at each location of cortex) found at baseline and at week 8.
Change from baseline in associations between motor measures and cortical thickness measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test) and MRI changes in cortical thickness (measured as the distance between the white and the pial surfaces at each location of cortex) found at baseline and at week 8.
Change from baseline in associations between self-report measures and cortical thickness measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number)) and MRI changes in cortical thickness (measured as the distance between the white and the pial surfaces at each location of cortex) found at baseline and at week 8.
Change from baseline in associations between motor performance and cortical thickness measures at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue) and MRI changes in cortical thickness (measured as the distance between the white and the pial surfaces at each location of cortex) found at baseline and at week 8.
Change from baseline in associations between cognitive and functional MRI task-based cortical activation at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test), and task-based functional MRI activation in the premotor cortex, the following contrasts will be calculated (Cued Tapping vs Rest) found at baseline and at week 8.
Change from baseline in associations between motor measures and functional MRI task-based cortical activation at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test) and task-based functional MRI activation in the premotor cortex, the following contrasts will be calculated (Cued Tapping vs Rest) found at baseline and at week 8.
Change from baseline in associations between self-report measures and functional MRI task-based cortical activation at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number)) and task-based functional MRI activation in the premotor cortex, the following contrasts will be calculated (Cued Tapping vs Rest) found at baseline and at week 8.
Change from baseline in associations between motor performance and functional MRI task-based cortical activation at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue) and task-based functional MRI activation in the premotor cortex, the following contrasts will be calculated (Cued Tapping vs Rest) found at baseline and at week 8.
Change from baseline in associations between cognitive and resting state fMRI connectivity in the auditory and sensorimotor networks measured at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test), and resting state connectivity will focus on nodes of auditory network and sensorimotor network strength in functional MRI activation at week 8 found at baseline and at week 8.
Change from baseline in associations between motor measures and resting-state fMRI connectivity in the auditory and sensorimotor networks measured at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test) and resting state connectivity will focus on nodes of auditory network and sensorimotor network strength in functional MRI activation at week 8 found at baseline and at week 8.
Change from baseline in associations between self-report measures and resting-state fMRI connectivity in the auditory and sensorimotor networks measured at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number)) and resting state connectivity will focus on nodes of auditory network and sensorimotor network strength in functional MRI activation at week 8 found at baseline and at week 8.
Change from baseline in associations between motor performance and resting-state fMRI connectivity in the auditory and sensorimotor networks measured at week 8. | Baseline and week 8
  Change in the strength of the associations (if any) between performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue) and resting state connectivity will focus on nodes of auditory network and sensorimotor network strength in functional MRI activation at week 8 found at baseline and at week 8.
Personality traits as predictor of interindividual differences in cognitive change from baseline to 8-week | Baseline and week 8
  Personality traits as measured by the Big Five-Short Form (administered at baseline) will be used as a covariate of changes from baseline to the 8-week timepoint in cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test).
Personality traits as predictor of interindividual differences in motor ability change from baseline to 8-week | Baseline and week 8
  Personality traits as measured by the Big Five-Short Form will be used as a covariate of changes from baseline to the 8-week timepoint in motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test).
Personality traits as predictor of interindividual differences in self-report measures from baseline to 8-week | Baseline and week 8
  Personality traits as measured by the Big Five-Short Form will be used as a covariate of changes from baseline to the 8-week timepoint in self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number))
Personality traits as predictor of interindividual differences in motor task performance from baseline to 8-week | Baseline and week 8
  Personality traits as measured by the Big Five-Short Form will be used as a covariate of changes from baseline to the 8-week timepoint in performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue).
Motivation to engage in musical activities as predictor of cognitive change from baseline to 8-week timepoint | Baseline and week 8
  We aim to assess the intrinsic motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) administered at the 8-week timepoint as a covariate of change from baseline to 8-week timepoint in cognitive measures (based on a composite score including scores from Digit Span Forward, Digit Span Backwards, Trail Making Test (inverted to indicate better outcome with higher number), Stroop Color Word Interference (inverted to indicate better outcome with higher number), Verbal Fluency Test, and the Rey Auditory Verbal-Learning Test).
Motivation to engage in musical activities as predictor of motor ability change from baseline to 8-week timepoint | Baseline and week 8
  We aim to assess the intrinsic motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) administered at the 8-week timepoint as a covariate of change from baseline to 8-week timepoint in motor measures (based on a composite score Grooved Pegboard Task (inverted to indicate better outcome with higher number), and Box and Blocks Test).
Motivation to engage in musical activities as predictor of self-report measures change from baseline to 8-week timepoint | Baseline and week 8
  We aim to assess the intrinsic motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) administered at the 8-week timepoint as a covariate of change from baseline to 8-week timepoint in self-report measures (based on a composite score of Quality of Life measure (inverted to indicate better outcome with higher number), and its visual analogue scale, Depression Anxiety Stress Scale (inverted to indicate better outcome with higher number)).
Motivation to engage in musical activities as predictor of motor task performance change from baseline to 8-week timepoint | Baseline and week 8
  We aim to assess the intrinsic motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) administered at the 8-week timepoint as a covariate of change from baseline to 8-week timepoint in performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue).
Motivation to engage in musical activities as predictor of change in resting-state connectivity of music-reward regions from baseline to 8-week timepoint | Baseline and week 8
  We seek to assess resting state connectivity in the nucleus accumbens (NAcc) with regions involved in music-reward as a proxy for motivation, namely superior temporal gyrus (STG), primary auditory cortex (A1), prefrontal cortex (PFC), the ventral striatum, and putamen while adding participant scores on the internal motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) as a covariate.
Motivation to engage in musical activities as predictor of change in white matter connectivity underlying music-reward regions from baseline to 8-week timepoint | Baseline and week 8
  We seek to assess changes in fractional anisotropy as measure of white matter integrity using diffuse tensor imaging (DTI) of white matter tracts underlying regions linked to music reward (NAcc, STG, A1, PFC, ventral striatum, and putamen). Namely, uncinate fasciculus, arcuate fasciculus, corpus callosum, cingulate bundle, fronto-occipital fasciculus, anterior limb of internal capsule, and the anterior thalamic radiation. Participant scores on a scale assessing the internal motivation to engage in musical activities using the Barcelona Music Reward Questionnaire (BMRQ) will be added as a covariate.
Musical background as a predictor of motor task performance change from baseline to 8-week timepoint | Baseline and week 8
  Musical background as assessed with the Goldsmith Musical Sophistication Index (GMSI) will be used as covariate in the change from baseline to 8-week timepoint in performance on the trained tasks (measured by a composite score of the number of correctly performed motor sequences and timing stability in synchrony with the onset of the cue).

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke E Hulst, PhD, Study Chair — Universiteit Leiden
Locations (1):
- Faculty of Social Science, Leiden University, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data relating to the main outcomes will be shared in online repository. Coded data will be published in an online scientific archive for the purpose of future research, in line with Open Science practices, and for the verification of findings for 10 years according to the Data Management Guidelines of the Health, Medical, and Neuropsychology Unit (v171220), Institute of Psychology, Faculty of Social and Behavioural Sciences at Leiden University. These data would not be traceable as they are not linked in any way to personal data. MRI data will be stored in the Open Science Framework (OSF) data repository and other platforms that may accommodate the large capacity of the data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Coded data will be published in online scientific archive without a time limit, all participant data, including physical documents will be archived at Faculty of Social and Behavioural Sciences at Leiden university for 10 years.
Access Criteria: Coded data that cannot be traceable to the participant identifying information will be published in an online repository, the web address of the repository will be included for each publication that results from the study. No restriction to access the publicly available data will be imposed, however, future studies that use the data of the study will be required to make reference to the study AND/OR the repository.

REFERENCES:
- [Background] Aloufi AE, Rowe FJ, Meyer GF. Behavioural performance improvement in visuomotor learning correlates with functional and microstructural brain changes. Neuroimage. 2021 Feb 15;227:117673. doi: 10.1016/j.neuroimage.2020.117673. Epub 2020 Dec 24. PMID 33359355
- [Background] Bermudez P, Lerch JP, Evans AC, Zatorre RJ. Neuroanatomical correlates of musicianship as revealed by cortical thickness and voxel-based morphometry. Cereb Cortex. 2009 Jul;19(7):1583-96. doi: 10.1093/cercor/bhn196. Epub 2008 Dec 10. PMID 19073623
- [Background] Blecher T, Tal I, Ben-Shachar M. White matter microstructural properties correlate with sensorimotor synchronization abilities. Neuroimage. 2016 Sep;138:1-12. doi: 10.1016/j.neuroimage.2016.05.022. Epub 2016 May 7. PMID 27165760
- [Background] Brown RM, Penhune VB. Efficacy of Auditory versus Motor Learning for Skilled and Novice Performers. J Cogn Neurosci. 2018 Nov;30(11):1657-1682. doi: 10.1162/jocn_a_01309. Epub 2018 Aug 29. PMID 30156505
- [Background] de Manzano O, Ullen F. Same Genes, Different Brains: Neuroanatomical Differences Between Monozygotic Twins Discordant for Musical Training. Cereb Cortex. 2018 Jan 1;28(1):387-394. doi: 10.1093/cercor/bhx299. PMID 29136105
- [Background] Chen JL, Rae C, Watkins KE. Learning to play a melody: an fMRI study examining the formation of auditory-motor associations. Neuroimage. 2012 Jan 16;59(2):1200-8. doi: 10.1016/j.neuroimage.2011.08.012. Epub 2011 Aug 16. PMID 21871571
- [Background] Chen JL, Zatorre RJ, Penhune VB. Interactions between auditory and dorsal premotor cortex during synchronization to musical rhythms. Neuroimage. 2006 Oct 1;32(4):1771-81. doi: 10.1016/j.neuroimage.2006.04.207. Epub 2006 Jun 14. PMID 16777432
- [Background] Denissen JJA, Geenen R, Soto CJ, John OP, van Aken MAG. The Big Five Inventory-2: Replication of Psychometric Properties in a Dutch Adaptation and First Evidence for the Discriminant Predictive Validity of the Facet Scales. J Pers Assess. 2020 May-Jun;102(3):309-324. doi: 10.1080/00223891.2018.1539004. Epub 2019 Jan 14. PMID 30638406
- [Background] EuroQol Research Foundation. (2019). EQ-5D-5L User Guide. https://euroqol.org/publications/user-guides/
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fine, E. M., & Delis, D. C. (2011). Delis-Kaplan Executive Functioning System. In J. S. Kreutzer, J. DeLuca, & B. Caplan (Eds.), Encyclopedia of Clinical Neuropsychology (pp. 796-801). Springer. https://doi.org/10.1007/978-0-387-79948-3_1539
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gaser C, Schlaug G. Brain structures differ between musicians and non-musicians. J Neurosci. 2003 Oct 8;23(27):9240-5. doi: 10.1523/JNEUROSCI.23-27-09240.2003. PMID 14534258
- [Background] Guo P, Li Q, Wang X, Li X, Wang S, Xie Y, Xie Y, Fu Z, Zhang X, Li S. Structural Covariance Changes of Anterior and Posterior Hippocampus During Musical Training in Young Adults. Front Neuroanat. 2020 May 19;14:20. doi: 10.3389/fnana.2020.00020. eCollection 2020. PMID 32508600
- [Background] Herholz SC, Coffey EB, Pantev C, Zatorre RJ. Dissociation of Neural Networks for Predisposition and for Training-Related Plasticity in Auditory-Motor Learning. Cereb Cortex. 2016 Jul;26(7):3125-34. doi: 10.1093/cercor/bhv138. Epub 2015 Jul 1. PMID 26139842
- [Background] Hudziak JJ, Albaugh MD, Ducharme S, Karama S, Spottswood M, Crehan E, Evans AC, Botteron KN; Brain Development Cooperative Group. Cortical thickness maturation and duration of music training: health-promoting activities shape brain development. J Am Acad Child Adolesc Psychiatry. 2014 Nov;53(11):1153-61, 1161.e1-2. doi: 10.1016/j.jaac.2014.06.015. Epub 2014 Sep 3. PMID 25440305
- [Background] Jenkinson M, Beckmann CF, Behrens TE, Woolrich MW, Smith SM. FSL. Neuroimage. 2012 Aug 15;62(2):782-90. doi: 10.1016/j.neuroimage.2011.09.015. Epub 2011 Sep 16. PMID 21979382
- [Background] Kissela BM, Khoury JC, Alwell K, Moomaw CJ, Woo D, Adeoye O, Flaherty ML, Khatri P, Ferioli S, De Los Rios La Rosa F, Broderick JP, Kleindorfer DO. Age at stroke: temporal trends in stroke incidence in a large, biracial population. Neurology. 2012 Oct 23;79(17):1781-7. doi: 10.1212/WNL.0b013e318270401d. Epub 2012 Oct 10. PMID 23054237
- [Background] Li Q, Wang X, Wang S, Xie Y, Li X, Xie Y, Li S. Musical training induces functional and structural auditory-motor network plasticity in young adults. Hum Brain Mapp. 2018 May;39(5):2098-2110. doi: 10.1002/hbm.23989. Epub 2018 Feb 5. PMID 29400420
- [Background] Lovibond, S. H., & Lovibond, P. F. (1995). Manual for the Depression Anxiety Stress Scales (2nd ed.). Psychology Foundation of Australia.
- [Background] Mas-Herrero, E., Marco-Pallares, J., Lorenzo-Seva, U., Zatorre, R. J., & Rodriguez-Fornells, A. (2013). Individual Differences in Music Reward Experiences. Music Perception, 31(2), 118-138. https://doi.org/10.1525/mp.2013.31.2.118
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Moore E, Schaefer RS, Bastin ME, Roberts N, Overy K. Diffusion tensor MRI tractography reveals increased fractional anisotropy (FA) in arcuate fasciculus following music-cued motor training. Brain Cogn. 2017 Aug;116:40-46. doi: 10.1016/j.bandc.2017.05.001. Epub 2017 Jun 12. PMID 28618361
- [Background] Müllensiefen, D., Gingras, B., Musil, J., & Stewart, L. (2014). Measuring the facets of musicality: The Goldsmiths Musical Sophistication Index (Gold-MSI). Personality and Individual Differences, 60, S35. https://doi.org/10.1016/j.paid.2013.07.081
- [Background] O'Callaghan G, O'Dowd A, Stapleton J, Merriman NA, Roudaia E, Newell FN. Changes in Regional Brain Grey-Matter Volume Following Successful Completion of a Sensori-Motor Intervention Targeted at Healthy and Fall-Prone Older Adults. Multisens Res. 2018 Jan 1;31(3-4):317-344. doi: 10.1163/22134808-00002604. PMID 31264622
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Pagano G, Ferrara N, Brooks DJ, Pavese N. Age at onset and Parkinson disease phenotype. Neurology. 2016 Apr 12;86(15):1400-1407. doi: 10.1212/WNL.0000000000002461. Epub 2016 Feb 10. PMID 26865518
- [Background] Rey, A. (1941). The psychological examination of cases of traumatic encephalopathy. 28, 286- 340.
- [Background] Rogge AK, Roder B, Zech A, Hotting K. Exercise-induced neuroplasticity: Balance training increases cortical thickness in visual and vestibular cortical regions. Neuroimage. 2018 Oct 1;179:471-479. doi: 10.1016/j.neuroimage.2018.06.065. Epub 2018 Jun 26. PMID 29959048
- [Background] Roy, E. A., & Square, P. A. (1994). CHAPTER 9-Neuropsychology of Movement Sequencing Disorders and Apraxia. In D. W. Zaidel (Ed.), Neuropsychology (pp. 183-218). Academic Press. https://doi.org/10.1016/B978-0-08-092668-1.50015-6
- [Background] Sachs ME, Ellis RJ, Schlaug G, Loui P. Brain connectivity reflects human aesthetic responses to music. Soc Cogn Affect Neurosci. 2016 Jun;11(6):884-91. doi: 10.1093/scan/nsw009. Epub 2016 Mar 10. PMID 26966157
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Background] Smith SM. Fast robust automated brain extraction. Hum Brain Mapp. 2002 Nov;17(3):143-55. doi: 10.1002/hbm.10062. PMID 12391568
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092
- [Background] Szameitat AJ, Schubert T, Muller HJ. How to test for dual-task-specific effects in brain imaging studies--an evaluation of potential analysis methods. Neuroimage. 2011 Feb 1;54(3):1765-73. doi: 10.1016/j.neuroimage.2010.07.069. Epub 2010 Aug 3. PMID 20688175
- [Background] Tavor I, Botvinik-Nezer R, Bernstein-Eliav M, Tsarfaty G, Assaf Y. Short-term plasticity following motor sequence learning revealed by diffusion magnetic resonance imaging. Hum Brain Mapp. 2020 Feb 1;41(2):442-452. doi: 10.1002/hbm.24814. Epub 2019 Oct 9. PMID 31596547
- [Background] Vaquero L, Ramos-Escobar N, Francois C, Penhune V, Rodriguez-Fornells A. White-matter structural connectivity predicts short-term melody and rhythm learning in non-musicians. Neuroimage. 2018 Nov 1;181:252-262. doi: 10.1016/j.neuroimage.2018.06.054. Epub 2018 Jun 19. PMID 29929006
- [Background] Wechsler, D. (2008). WAIS-IV: Wechsler Adult Intelligence Scale-Fourth Edition (4th ed.). Pearson.
- [Background] Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proc Natl Acad Sci U S A. 2000 Sep 26;97(20):11050-5. doi: 10.1073/pnas.200033797. PMID 10984517
- [Background] Mas-Herrero E, Dagher A, Farres-Franch M, Zatorre RJ. Unraveling the Temporal Dynamics of Reward Signals in Music-Induced Pleasure with TMS. J Neurosci. 2021 Apr 28;41(17):3889-3899. doi: 10.1523/JNEUROSCI.0727-20.2020. Epub 2021 Mar 29. PMID 33782048
- [Background] Gold BP, Mas-Herrero E, Zeighami Y, Benovoy M, Dagher A, Zatorre RJ. Musical reward prediction errors engage the nucleus accumbens and motivate learning. Proc Natl Acad Sci U S A. 2019 Feb 19;116(8):3310-3315. doi: 10.1073/pnas.1809855116. Epub 2019 Feb 6. PMID 30728301
- [Background] Belfi AM, Loui P. Musical anhedonia and rewards of music listening: current advances and a proposed model. Ann N Y Acad Sci. 2020 Mar;1464(1):99-114. doi: 10.1111/nyas.14241. Epub 2019 Sep 23. PMID 31549425
- [Background] Koch K, Wagner G, Schachtzabel C, Schultz CC, Gullmar D, Reichenbach JR, Sauer H, Zimmer C, Schlosser RG. Association between white matter fiber structure and reward-related reactivity of the ventral striatum. Hum Brain Mapp. 2014 Apr;35(4):1469-76. doi: 10.1002/hbm.22284. Epub 2013 Apr 24. PMID 23616433
- [Background] Mas-Herrero E, Maini L, Sescousse G, Zatorre RJ. Common and distinct neural correlates of music and food-induced pleasure: A coordinate-based meta-analysis of neuroimaging studies. Neurosci Biobehav Rev. 2021 Apr;123:61-71. doi: 10.1016/j.neubiorev.2020.12.008. Epub 2021 Jan 10. PMID 33440196
- [Background] Shany O, Singer N, Gold BP, Jacoby N, Tarrasch R, Hendler T, Granot R. Surprise-related activation in the nucleus accumbens interacts with music-induced pleasantness. Soc Cogn Affect Neurosci. 2019 May 17;14(4):459-470. doi: 10.1093/scan/nsz019. PMID 30892654